CLINICAL TRIAL: NCT06798025
Title: Comparative Study Between Three Different Modalities for Treatment of Inflammatory Punctal Stenosis
Brief Title: Three Different Modalities for Treatment of Inflammatory Punctal Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Yomna EL-Saied Mohamed Ibrahim, Resident of Ophthalmology, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36264MS245/2/23
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Modalities; Treatment; Inflammatory Punctal Stenosis
MeSH Terms: interventions — Dosage Forms; Triamcinolone Acetonide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Patients were treated with punctal dilatation only
  Interventions: Procedure: Punctal dilation
- Group B (Experimental): Patients were treated with a combination of punctual dilation and topical medication in the form of preservative-free steroid eye drops based on dexamethasone sodium phosphate (0.1%) and preservative-free artificial tears based on sodium hyaluronate, polyethylene, and propylene Glycol.
  Interventions: Drug: Punctal dilation and topical medication
- Group C (Experimental): Patients were treated with a peri-punctual injection of Triamcinolone acetonide.
  Interventions: Drug: Triamcinolone acetonide

INTERVENTIONS:
Procedure: Punctal dilation — Patients were treated with punctal dilatation only.
  Arms: Group A
Drug: Punctal dilation and topical medication — Patients were treated with a combination of punctal dilation and topical medication in the form of preservative-free steroid eye drops based on dexamethasone sodium phosphate (0.1%) and preservative-free artificial tears based on sodium hyaluronate, polyethylene, and propylene Glycol.
  Arms: Group B
Drug: Triamcinolone acetonide — Patients were treated with a peri-punctual injection of Triamcinolone acetonide.
  Arms: Group C

SUMMARY:
This study aimed to compare the efficacy of three various modalities of treatment of inflammatory punctal stenosis (Punctal dilatation alone, combined punctal dilatation with topical medications, or peri-punctal injection of Triamcinolone acetonide)

DETAILED DESCRIPTION:
Acquired punctal stenosis is a condition in which the external opening of the lacrimal canaliculus, located in the nasal part of the palpebral margin, is narrowed or occluded. This condition results from chronic inflammation of the external punctum, leading to gradual fibrotic changes in the ostium, followed by progressive occlusion of the duct.

Different modalities were described for the treatment of acquired punctual stenosis. Repeated dilatation of the stenotic punctum is a simple procedure that may provide temporary improvement of the symptoms, but restenosis is common unless additional procedures are performed. Many other methods were used to augment punctual size, including 1-snip, 2-snip, and 3-snip punctoplasty, supplemented with adding sutures or Mini-Monoka insertion and punch punctoplasty.

ELIGIBILITY:
Inclusion Criteria:

* Age from 33 to 75.
* Both sexes.
* Patients with inflammatory punctal stenosis or occlusion complaining of symptomatic epiphora.

Exclusion Criteria:

* Subjects with previous lacrimal surgeries.
* Subjects with lid margin malposition such as ectropion, entropion, or lid retraction.
* Subjects with medial lid masses obscuring the punctum.
* Subjects with a history of ocular trauma involving the medial aspect of the lid margin.

Ages: 33 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Degree of patient satisfaction | 3 months postoperatively
  The degree of patient satisfaction was assessed using 3-point Likert Scale (1=Not satisfied, 2: No Difference, 3:Satisfied)

SECONDARY OUTCOMES:
Punctal diameter | 3 months postoperatively
  The punctal diameter of cases was measured before and after 1 month and 3 months of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.